CLINICAL TRIAL: NCT03205722
Title: The Effectiveness of Nivolumab (OPDIVO®) Monotherapy as First-Line Therapy in Adults With Advanced (Unresectable or Metastatic) Melanoma: An Early Retrospective, Observational Study in Germany
Brief Title: The Effectiveness of Nivolumab Monotherapy as First-Line Therapy in Adults With Advanced Melanoma in Germany
Status: Withdrawn | Type: Observational
Why Stopped: Business objectives have changed
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-939
Record Dates: First submitted 2017-06-29; First posted 2017-07-02 (Actual); Last update posted 2018-04-09 (Actual); Status verified 2018-04

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Melanoma patients with 1st-line Nivo treatment: Non-Interventional. Patients with advanced melanoma treated with nivolumab monotherapy prescribed as first-line therapy between June 2015 and June 2016.
  Interventions: Other: Non-Interventional

INTERVENTIONS:
Other: Non-Interventional — Non-Interventional

SUMMARY:
A retrospective, observational study based on chart reviews for patients with advanced melanoma treated with nivolumab monotherapy prescribed as first-line therapy between June 2015 and June 2016, conducted in a representative sample of sites in Germany.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with a primary diagnosis of advanced melanoma (histologically confirmed stage III [unresectable] or stage IV skin, ocular, or mucosal melanoma)
* Newly initiated with nivolumab monotherapy as their first-line therapy for previously untreated advanced melanoma between June 2015 and June 2016
* At least 18 years of age at time of treatment decision

Exclusion Criteria:

* Patients with a current primary diagnosis of a cancer other than advanced melanoma ie, a cancer other than melanoma that requires systemic or other treatment
* Patients currently included in an interventional clinical trial for his/her locally advanced or metastatic melanoma. Patients who have completed their participation in an interventional trial; or who are not receiving study drug anymore and who are only followed-up for overall survival can be enrolled. In case of a blinded study, the treatment arm (ie, type of administered treatment) needs to be known.
* Patients < 18 years of age at time of treatment initiation

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients diagnosed with advanced melanoma who were initiated with nivolumab monotherapy as their first-line therapy in Germany between June 2015 and June 2016.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-01-05 (Estimated); Primary Completion 2018-07-30 (Estimated); Study Completion 2018-07-30 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | Approximately 23 months
  OS for adult patients with advanced (unresectable or metastatic) melanoma treated with nivolumab monotherapy as first-line therapy from date of advanced diagnosis, and from the start of treatment with nivolumab over the first 23 months after treatment initiation, overall.

SECONDARY OUTCOMES:
OS from date of advanced diagnosis | Approximately 23 months
progression-free survival (PFS) | Approximately 23 months
best overall response rate (BORR) | Approximately 23 months
best overall response (BOR) | Approximately 23 months
Distribution of Best Overall Response (BOR) by Severity of melanoma at initiation of treatment | Approximately 23 months
Best Overall Response (BOR) in patients greater than or equal to 65 years old | Approximately 23 months
Best Overall Response (BOR) in Eastern Cooperative Oncology Group (ECOG) performance status greater than or equal to 2 | Approximately 23 months
Distribution of Best Overall Response (BOR) by Mutational status | Approximately 23 months
Best Overall Response (BOR) in Patients with brain metastases | Approximately 23 months
Distribution of Best Overall Response (BOR) by Melanoma subtype | Approximately 23 months
Distribution of incidence of Adverse Events (AEs) | Approximately 23 months
Distribution of severity of Adverse Events (AEs) | Approximately 23 months
Distribution of management of Adverse Events (AEs) | Approximately 23 months
Distribution of socio-demographic characteristics in adult patients with advanced melanoma treated with nivolumab monotherapy as first-line therapy | Approximately 23 months
  Socio-demographic characteristics (Gender, Height, Weight, Age) will be summarized using descriptive statistics
Distribution of clinical characteristics in adult patients with advanced melanoma treated with nivolumab monotherapy as first-line therapy | Approximately 23 months
  Clinical characteristics (Initial Diagnosis of melanoma, Histological subtypes, Performance status, Comorbidities, history of cancer) will be summarized using descriptive statistics
Distribution of Treatment Patterns | Approximately 23 months
  Details on Prior and Evolution of Current Treatment Patterns will be summarized using descriptive statistics.
Distribution of Healthcare Resource Utilization | Approximately 23 months
  Healthcare Resource Utilization will be summarized using descriptive statistics
Duration of nivolumab treatment | Approximately 23 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx